CLINICAL TRIAL: NCT02437084
Title: Relationship Between Insulin Resistance and Statin Induced Type 2 Diabetes, and Integrative Personal Omics Profiling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Joshua Knowles, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STANFORD
Record Dates: First submitted 2015-04-24; First posted 2015-05-07 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Hyperlipidemia; Insulin Resistance; Type 2 Diabetes
Keywords: statin; diabetes; insulin resistance; insulin secretion
MeSH Terms: conditions — Hyperlipidemias; Insulin Resistance; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individuals without diabetes eligible to receive statin therapy (Other): Eligible participants will receive 40 mg of atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Study subjects will receive atorvastatin 40 mg for 10 weeks.
  Other Names: Lipitor

SUMMARY:
Background:

There is general agreement that statin-treatment of patients to lower plasma cholesterol levels can increase the incidence of type 2 diabetes mellitus (T2D) in some individuals1-5. The physiologic mechanism for the increased risk for T2D from statin treatment is unknown but could result from effects on insulin sensitivity or insulin secretion. This study will evaluate how the medication atorvastatin (trade name Lipitor) works in non-diabetic individuals in regards to its effect on insulin sensitivity and insulin secretion to help further understand the possible cause of the increased occurrence of T2D in people who are at risk for T2D. This research study will also examine what metabolic characteristics and variables (for example insulin resistance, high triglycerides, or both) will identify those people at highest risk of statin-induced T2D.

The goals of this study are to:

1. determine the effect of high-intensity atorvastatin (40 mg/day) for ~ 10 weeks on insulin sensitivity and insulin secretion (defined with gold standard methods) (PRIMARY OUTCOMES) as well as other glycemic traits (SECONDARY OUTCOMES);
2. compare a number of cardio-metabolic characteristics (e.g. weight, lipids) before, during, and after administration of atorvastatin;
3. determine if significant deterioration of insulin action and/or secretion following statin treatment will be confined to those with baseline insulin resistance (PRE-SPECIFIED SUBGROUP ANALYSES);
4. perform Personal Omics Profiling (iPOP) 6,7 before and after taking atorvastatin to examine treatment-associated changes in all baseline variables and to analyze not only previously-known drug efficacy but also untargeted drug efficacy (EXPLORATORY ANALYSES).

General approach:

This will be an open-label study to evaluate the diabetogenic effect of atorvastatin (40 mg/day for 10 weeks) on both insulin action and insulin secretion in nondiabetic individuals. To ensure we recruit individuals across a broad range of insulin sensitivity, we will target recruitment to enrich for those with combined increases in LDL-C and TG concentrations (see SIGNIFICANCE and RATIONALE). The experimental population will consist of ~75 apparently healthy, non-diabetic volunteers eligible for statin therapy but without pre-existing atherosclerotic cardiovascular disease. Following baseline assessments of co-primary outcome measures: insulin sensitivity (by insulin suppression test, IST) and insulin secretion (by graded glucose infusion test, GGIT), participants will be placed on a weight maintenance diet and treated with 40 mg/day of atorvastatin. All baseline measurements will be repeated ~10 weeks later with iPOP8 measurements done at baseline, at weeks 2, 4, and 10 on atorvastatin, and at weeks 4 and 8 off atorvastatin.

DETAILED DESCRIPTION:
1. SIGNIFICANCE

   Statins and the risk of T2D: Statin treatment is associated with an increase in incident T2D.1-4 5

   Mechanism of statin-induced T2D: It is unclear whether statins increase the risk of T2D by decreasing insulin action, secretion, or both. Several manuscripts have been published that substantially increase understanding of the link between statin use and incident T2D. Swerdlow, et al.2 based on evidence from genetic analysis and randomized trials, concluded that the increased risk of T2D noted with statins is at least "partially explained by HMG-coenzyme A reductase (HMGCR) inhibition." They also noted an association of weight gain with HMGCR variants in statin-treated patients, leading to the notion that decreases in insulin sensitivity contribute to statin-induced diabetes. In that context, Cederberg, at al.9 have shown in a large prospective study (n=8749 men) that participants treated with statins (n=2142) had a 46% increase in incident T2D, associated with a 24% decrease in insulin sensitivity and a 12% decrease in insulin secretion assessed by surrogate measures.

   Identifying those with at enhanced risk of statin-induced T2D: Studies of 3 randomized clinical trials with atorvastatin by David Waters' group 1,3,4 have demonstrated that "baseline fasting glucose, body mass index, hypertension, and fasting triglycerides were independent predictors of T2D." These abnormalities form a cluster attributed to insulin resistance.10 Since insulin resistance is a predictor of developing T2D, it seems likely that the more insulin resistant the individuals are before treatment, the greater is their risk to for statin-induced T2D.

   In that context, relatively little attention has been given to the role that metabolic heterogeneity in patients with elevated LDL-C concentrations might play in statin-induced T2D. Specifically, subjects with elevated LDL-C concentrations, whose plasma triglyceride (TG) concentrations are also elevated, are insulin resistant, hyperinsulinemic, and glucose intolerant as compared to those with isolated LDL-C levels. As such, this subset of patients with elevated LDL-C concentrations can be viewed as being at a "tipping point," and any adverse effect of statins on insulin action and/or secretion, irrespective of how mediated, places them at enhanced risk to develop statin-induced diabetes. Indeed, we have shown (Kohli et al)1 that patients with both insulin resistance (as estimated by high TGs) and prediabetes are at particularly high risk of statin-induced T2D.

   We seek to address 2 important unanswered questions: Do statins primarily affect insulin resistance or insulin secretion?; Are there subsets of individuals at highest risk of statin-induced T2D?
2. RATIONALE, HYPOTHESIS

   Rationale:

   T2D develops when insulin resistant individuals cannot maintain the degree of compensatory hyperinsulinemia needed to maintain normal glucose tolerance. However, significant fundamental questions remain. For example, what is the cellular/molecular link between statin treatment and changes in insulin action and secretion?

   This proposal is based on the premise that studying the effect of statins on insulin action and insulin secretion using "gold standard" methods will help determine if statins adversely affect the risk of T2D by increasing insulin resistance or decreasing insulin secretion. We use the insulin suppression test (with the read-out of steady-state plasma glucose, SSPG) to ascertain insulin sensitivity and the graded glucose infusion test (with the readout of insulin secretion rate, ISR) to ascertain insulin secretion both before and after statin treatment in non-diabetic individuals.

   We hypothesize that treatment with atorvastatin 40 mg/day for approximately 10 weeks will impair insulin sensitivity and/or insulin secretion and that this effect may be exacerbated in those with underlying insulin resistance. Thus, we plan to look at the effect of atorvastatin not only in all participants but also in subsets of individuals with baseline insulin resistance (which will be enriched for by recruiting volunteers with elevated plasma TG levels (≥150 mg/dL) at baseline. The rationale for this is that plasma TGs are a surrogate measure for insulin resistance with a modest correlation with the direct measure of insulin resistance (steady-state plasma glucose) measured by the insulin suppression test. Clinically, subjects with elevated TGs prior to statin treatment would have substantial clinical benefit from statins, and one of investigators' secondary goals is to demonstrate that a simple measurement of plasma TG concentration (as a surrogate for insulin resistance) can help identify those most at risk of statin induced derangements in glycemic control. Consequently, we propose to enroll nondiabetic volunteers at high-risk for T2D, free of known atherosclerotic cardiovascular disease (ASCVD), not receiving statins, eligible for statin therapy according to ACC/AHA (American College for Cardiology/American Heart Association) 2013 guidelines.11 We will also target recruitment efforts to enrich for subjects with plasma TG concentration ≥ 150 mg/dL to ensure that we enroll subjects across the range of insulin sensitivity.

   Hypothesis: We hypothesize that high intensity atorvastatin treatment for approximately 10 weeks will impair insulin sensitivity and/or insulin secretion and that this effect may be exacerbated in those with underlying insulin resistance.
3. STUDY DESIGN

   Sample Size

   • We aim to recruit and retain 75 total participants in this study.

   Study Location

   • Clinical and Translational Research Unit (CTRU) at 800 Welch Road, Palo Alto, CA 94304.

   Duration

   • We anticipate that the entire study will take 4 - 5 years through the end of data analysis. Each eligible candidate who voluntarily consents to participate in the study will be active in the study for a total of 5 months from screening to the end of their last visit.
4. STUDY PROCEDURES

   Recruitment

   Preliminary recruitment strategies will include:

   Volunteers will be recruited from the San Francisco Bay Area through advertisements in newspapers, posted flyers, and the social networking site NextDoor as well as from the Preventive Cardiology Clinics at Stanford Health Care. Our goal is to ensure recruitment across a broad range of insulin sensitivity. Prior work from our group and others has shown that high plasma TG concentrations are associated with increased insulin resistance as assessed by reference measures. Therefore, we will target advertisements to enrich for individuals with high TG levels (> 150 mg/dL) as a surrogate for increased insulin resistance.

   Participant Visits and Procedures

   Potential participants will be screened initially when they call or email in response to recruitment ads, or a letter from their MD, describing the study as follows:

   Preliminary intake will occur over the phone.

   Visit 1 Screening visit.

   Visit 2: Oral Glucose Tolerance Test (OGTT): This test will take approximately 3 hours.

   i) Glycemic status: Participants will be classified as having normal glucose tolerance (NGT), isolated impaired fasting glucose (IFG), isolated impaired glucose tolerance (IGT), or combined IFG/IGT12. In addition, the total integrated plasma glucose response during the OGTT will be calculated by the trapezoidal method (Glucose-AUC).

   ii) β-cell function: Calculations of the Insulin Secretion- Sensitivity Index-2 (ISSI-2) will be used to quantify insulin secretory function 13, if for some reason a graded glucose infusion study is not done. The ISSI-2 is a validated OGTT- derived method to measure of β-cell function, analogous to the disposition index obtained from the intravenous glucose tolerance test 14. It is calculated by multiplying the insulin secretory response during the OGTT (Insulin-AUC/Glucose-AUC) by insulin resistance (Matsuda index).

   The fasting and 2-hour glucose results will be discussed with the study participant and a copy of the results will be given to them.

   Visit 3. Graded Glucose Infusion, GGIT 15,16: This test will take approximately 6 hours.

   This test is designed to assess the ability of the pancreas to produce insulin in response to a graded glucose infusion. During this test, subjects will have two small IV catheters placed, one in each arm. One IV will be used for drawing samples and the other for the infusion of glucose. During the GGIT, continuous intravenous infusions of glucose will be given at progressively increasing rates: 1, 2, 3, 4, 5, 6, and 8 kg/min in six infusion periods of 40-min duration. Blood samples will be collected for measurements of glucose, insulin, and C-peptide concentrations at fasting and at 30 min and 40 min into each infusion period. The two values during the last 10 min of each infusion period will be averaged. The amount of blood taken for this test will 47.5 ml.

   Visit 4.Insulin Suppression test, IST 17,18: This test will take approximately 6 hours.

   This test is designed to determine whole body insulin sensitivity. Following an overnight fast, subjects will have an IV placed in each arm. One for collection of blood and the other for infusion with octreotide (0.27 μg/m2/min), insulin (32 mU/m2/min), and glucose (267 mg/m2/min) for 180 minutes. During the test, endogenous insulin is suppressed and all individuals are given the same concentration of insulin, based on their body surface area. Blood is drawn every 30 minutes for 150 minutes and then at 10-minute intervals from 150 to 180 minutes of the infusion to measure plasma glucose and insulin concentrations. The mean of the last four values is used as the steady-state plasma insulin (SSPI) and glucose (SSPG) concentrations for each individual. As SSPI concentrations are similar in all subjects during the IST, the SSPG concentration provides a direct measure of the ability of insulin to mediate disposal of an infused glucose load; the higher the SSPG concentration, the more insulin resistant the individual. Labs to check kidney and liver function plus a lipid panel and a urine pregnancy test (if appropriate) will be done at this visit. Blood drawn or IST will be 58.5 ml and 5 ml for SHC labs.

   Labs for iPOP will be drawn at this time and additional samples will be obtained for transcriptome, microbiome, metabolome, and proteome analysis in blood; nasal, tongue, skin surface swabs; urine; and stool.

   The study drug, atorvastatin 40 mg will be given to study participants, once all labs have been reviewed and participant qualifies.

   Visit 5-7: Visits will be every 2 weeks for a total of 10 weeks on study medication (statin). Participants will be assessed for any side effects or adverse events (AE) on the statin. Adherence to study medication will be assessed at each visit.

   Visit 8: Weight, vital signs, and OGTT described above.

   Visit 9: Repeat GGIT as described above.

   Visit 10: Repeat IST and iPOP lab testing and samples as described above. At the end of this visit, the statin will be stopped and the study participant would be scheduled for 4- and 8-week follow up visits.

   Visit 11: One month off statin study visit - weight, vital signs, and iPOP laboratory testing and samples will be done as described above.

   Visit 12: Last study visit - weight, vital signs, and iPOP laboratory testing and samples will be done as described above.

   Participants will be asked to fill out questionnaire about her/his physical activity status, food and eating habits, and stress at the time of each iPOP.
5. STATISTICAL CONSIDERATIONS

Based on our prior work19, we calculated that with 60 subjects, we would be able to detect an 8% change in SSPG concentration and an 8% change in ISRAUC after atorvastatin therapy with 80% power and two-side significance level of 5% using a paired samples t test. Thus, we estimated needing to enroll 75 subjects with an anticipated a dropout rate of 20%.

Summary statistics will be reported as median (interquartile range) or number (percent) of participants unless otherwise specified. Shapiro-Wilk tests will be used to assess normality of data, and variables that are not normally distributed will be log-transformed. Percent changes in variables will be calculated by the formula: [(end-of study value) - (baseline value) / baseline value] x 100. Paired samples t tests will be used to compare baseline and end-of-study means. One sample t tests will be employed to evaluate whether percent changes in variables are significantly different from zero (no change). Pearson correlation coefficients will be calculated to determine the strength of association between variables of interest. Prespecified subgroup analyses will be carried out by stratifying for insulin resistant versus insulin sensitive subjects. The SSPG concentration median will be used to define subjects as being insulin resistant or insulin sensitive. Insulin resistant and insulin sensitive group means will be compared by independent sample t tests and proportions by chi-square tests or Fisher's exact tests. Statistical analyses will be performed by using statistical software IBM SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 30 - 70 years old
2. BMI: 20 - 37 kg/m2
3. Without diabetes as defined by fasting plasma glucose <126 mg/dL and not taking glucose lowering medications
4. Eligible for statin therapy for primary prevention of ASCVD based on LDL-C ≥ 130 mg/dL, > 5% ASCVD risk over 10 years, or hs-CRP ≥ 2.0 mg/L

Exclusion Criteria:

1. Younger than 30 or older than 70 years
2. Persons with any significant co-morbidities, such as diabetes (fasting glucose ≥ 126 mg/dL or use of glucose lowering medications), active coronary artery disease, heart failure, accelerated or malignant hypertension, kidney disease (creatinine ≥ 1.5 mg/dL), liver disease (alanine aminotransferase > 2 times upper limit of normal), or severe anemia (hematocrit < 30%).
3. Individuals taking any medications for weight loss or known to influence insulin sensitivity.
4. Pregnant or lactating
5. Women unwilling to use an effective birth control method
6. History of statin intolerance

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Knowles, M.D. Ph. D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohli P, Knowles JW, Sarraju A, Waters DD, Reaven G. Metabolic Markers to Predict Incident Diabetes Mellitus in Statin-Treated Patients (from the Treating to New Targets and the Stroke Prevention by Aggressive Reduction in Cholesterol Levels Trials). Am J Cardiol. 2016 Nov 1;118(9):1275-1281. doi: 10.1016/j.amjcard.2016.07.054. Epub 2016 Aug 12. PMID 27614854
- [Background] Swerdlow DI, Preiss D, Kuchenbaecker KB, Holmes MV, Engmann JE, Shah T, Sofat R, Stender S, Johnson PC, Scott RA, Leusink M, Verweij N, Sharp SJ, Guo Y, Giambartolomei C, Chung C, Peasey A, Amuzu A, Li K, Palmen J, Howard P, Cooper JA, Drenos F, Li YR, Lowe G, Gallacher J, Stewart MC, Tzoulaki I, Buxbaum SG, van der A DL, Forouhi NG, Onland-Moret NC, van der Schouw YT, Schnabel RB, Hubacek JA, Kubinova R, Baceviciene M, Tamosiunas A, Pajak A, Topor-Madry R, Stepaniak U, Malyutina S, Baldassarre D, Sennblad B, Tremoli E, de Faire U, Veglia F, Ford I, Jukema JW, Westendorp RG, de Borst GJ, de Jong PA, Algra A, Spiering W, Maitland-van der Zee AH, Klungel OH, de Boer A, Doevendans PA, Eaton CB, Robinson JG, Duggan D; DIAGRAM Consortium; MAGIC Consortium; InterAct Consortium; Kjekshus J, Downs JR, Gotto AM, Keech AC, Marchioli R, Tognoni G, Sever PS, Poulter NR, Waters DD, Pedersen TR, Amarenco P, Nakamura H, McMurray JJ, Lewsey JD, Chasman DI, Ridker PM, Maggioni AP, Tavazzi L, Ray KK, Seshasai SR, Manson JE, Price JF, Whincup PH, Morris RW, Lawlor DA, Smith GD, Ben-Shlomo Y, Schreiner PJ, Fornage M, Siscovick DS, Cushman M, Kumari M, Wareham NJ, Verschuren WM, Redline S, Patel SR, Whittaker JC, Hamsten A, Delaney JA, Dale C, Gaunt TR, Wong A, Kuh D, Hardy R, Kathiresan S, Castillo BA, van der Harst P, Brunner EJ, Tybjaerg-Hansen A, Marmot MG, Krauss RM, Tsai M, Coresh J, Hoogeveen RC, Psaty BM, Lange LA, Hakonarson H, Dudbridge F, Humphries SE, Talmud PJ, Kivimaki M, Timpson NJ, Langenberg C, Asselbergs FW, Voevoda M, Bobak M, Pikhart H, Wilson JG, Reiner AP, Keating BJ, Hingorani AD, Sattar N. HMG-coenzyme A reductase inhibition, type 2 diabetes, and bodyweight: evidence from genetic analysis and randomised trials. Lancet. 2015 Jan 24;385(9965):351-61. doi: 10.1016/S0140-6736(14)61183-1. Epub 2014 Sep 24. PMID 25262344
- [Background] Kohli P, Waters DD, Nemr R, Arsenault BJ, Messig M, DeMicco DA, Laskey R, Kastelein JJP. Risk of new-onset diabetes and cardiovascular risk reduction from high-dose statin therapy in pre-diabetics and non-pre-diabetics: an analysis from TNT and IDEAL. J Am Coll Cardiol. 2015 Feb 3;65(4):402-404. doi: 10.1016/j.jacc.2014.10.053. No abstract available. PMID 25634843
- [Background] Waters DD, Ho JE, Boekholdt SM, DeMicco DA, Kastelein JJ, Messig M, Breazna A, Pedersen TR. Cardiovascular event reduction versus new-onset diabetes during atorvastatin therapy: effect of baseline risk factors for diabetes. J Am Coll Cardiol. 2013 Jan 15;61(2):148-52. doi: 10.1016/j.jacc.2012.09.042. Epub 2012 Dec 5. PMID 23219296
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Li-Pook-Than J, Snyder M. iPOP goes the world: integrated personalized Omics profiling and the road toward improved health care. Chem Biol. 2013 May 23;20(5):660-6. doi: 10.1016/j.chembiol.2013.05.001. PMID 23706632
- [Background] Snyder M. iPOP and its role in participatory medicine. Genome Med. 2014 Jan 30;6(1):6. doi: 10.1186/gm512. eCollection 2014. PMID 24479626
- [Background] Chen R, Mias GI, Li-Pook-Than J, Jiang L, Lam HY, Chen R, Miriami E, Karczewski KJ, Hariharan M, Dewey FE, Cheng Y, Clark MJ, Im H, Habegger L, Balasubramanian S, O'Huallachain M, Dudley JT, Hillenmeyer S, Haraksingh R, Sharon D, Euskirchen G, Lacroute P, Bettinger K, Boyle AP, Kasowski M, Grubert F, Seki S, Garcia M, Whirl-Carrillo M, Gallardo M, Blasco MA, Greenberg PL, Snyder P, Klein TE, Altman RB, Butte AJ, Ashley EA, Gerstein M, Nadeau KC, Tang H, Snyder M. Personal omics profiling reveals dynamic molecular and medical phenotypes. Cell. 2012 Mar 16;148(6):1293-307. doi: 10.1016/j.cell.2012.02.009. PMID 22424236
- [Background] Cederberg H, Stancakova A, Yaluri N, Modi S, Kuusisto J, Laakso M. Increased risk of diabetes with statin treatment is associated with impaired insulin sensitivity and insulin secretion: a 6 year follow-up study of the METSIM cohort. Diabetologia. 2015 May;58(5):1109-17. doi: 10.1007/s00125-015-3528-5. Epub 2015 Mar 10. PMID 25754552
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S14-S31. doi: 10.2337/dc20-S002. PMID 31862745
- [Background] Retnakaran R, Shen S, Hanley AJ, Vuksan V, Hamilton JK, Zinman B. Hyperbolic relationship between insulin secretion and sensitivity on oral glucose tolerance test. Obesity (Silver Spring). 2008 Aug;16(8):1901-7. doi: 10.1038/oby.2008.307. Epub 2008 Jun 12. PMID 18551118
- [Background] Weyer C, Bogardus C, Mott DM, Pratley RE. The natural history of insulin secretory dysfunction and insulin resistance in the pathogenesis of type 2 diabetes mellitus. J Clin Invest. 1999 Sep;104(6):787-94. doi: 10.1172/JCI7231. PMID 10491414
- [Background] Jones CN, Pei D, Staris P, Polonsky KS, Chen YD, Reaven GM. Alterations in the glucose-stimulated insulin secretory dose-response curve and in insulin clearance in nondiabetic insulin-resistant individuals. J Clin Endocrinol Metab. 1997 Jun;82(6):1834-8. doi: 10.1210/jcem.82.6.3979. PMID 9177392
- [Background] Kim SH, Abbasi F, Chu JW, McLaughlin TL, Lamendola C, Polonsky KS, Reaven GM. Rosiglitazone reduces glucose-stimulated insulin secretion rate and increases insulin clearance in nondiabetic, insulin-resistant individuals. Diabetes. 2005 Aug;54(8):2447-52. doi: 10.2337/diabetes.54.8.2447. PMID 16046313
- [Background] Shen SW, Reaven GM, Farquhar JW. Comparison of impedance to insulin-mediated glucose uptake in normal subjects and in subjects with latent diabetes. J Clin Invest. 1970 Dec;49(12):2151-60. doi: 10.1172/JCI106433. PMID 5480843
- [Background] Pei D, Jones CN, Bhargava R, Chen YD, Reaven GM. Evaluation of octreotide to assess insulin-mediated glucose disposal by the insulin suppression test. Diabetologia. 1994 Aug;37(8):843-5. doi: 10.1007/BF00404344. No abstract available. PMID 7988789
- [Background] Kim SH, Liu A, Ariel D, Abbasi F, Lamendola C, Grove K, Tomasso V, Reaven G. Pancreatic beta cell function following liraglutide-augmented weight loss in individuals with prediabetes: analysis of a randomised, placebo-controlled study. Diabetologia. 2014 Mar;57(3):455-62. doi: 10.1007/s00125-013-3134-3. Epub 2013 Dec 11. PMID 24326527
- [Derived] Abbasi F, Lamendola C, Harris CS, Harris V, Tsai MS, Tripathi P, Abbas F, Reaven GM, Reaven PD, Snyder MP, Kim SH, Knowles JW. Statins Are Associated With Increased Insulin Resistance and Secretion. Arterioscler Thromb Vasc Biol. 2021 Nov;41(11):2786-2797. doi: 10.1161/ATVBAHA.121.316159. Epub 2021 Aug 26. PMID 34433298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed between 2015 and 2019 at the Stanford Clinical and Translational Research Unit. Volunteers were recruited from the San Francisco Bay Area through advertisements in newspapers, posted flyers, the social networking site NextDoor and the Preventive Cardiology Clinics at Stanford Health Care.
Pre-assignment Details: Of the 115 participants enrolled, 40 declined to participate and 75 started treatment with atorvastatin 40 mg daily. Individuals who were receiving statin therapy at the time of enrollment underwent a 4-week statin washout with approval of their treating physician.
Groups:
- Atorvastatin Treatment: Participants received treatment with atorvastatin 40 mg daily for 10 weeks.
Period: Overall Study
Arm/Group | Atorvastatin Treatment
Started | 75
Completed | 72
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed both baseline and end-of-study tests and did not receive treatment with a corticosteroid.
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 50
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 71
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 27.8 [24.8 to 30.7]

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Plasma Glucose (SSPG)
Description: Insulin sensitivity measured by SSPG concentration (mg/dL) during the insulin suppression test.
Time Frame: baseline, week 9 or 10
Population: Participants who completed both baseline and end-of-study insulin suppression tests and did not receive treatment with a corticosteroid.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 70
mg/dL
  Baseline | 130 [85 to 193]
  End of Study | 139 [93 to 211]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in steady-state plasma glucose (SSPG) concentration after treatment with atorvastatin 40 mg daily for 9 - 10 weeks; Test type: Other; p = 0.01, Paired samples t test, 2 sided; SSPG concentration was log-transformed for statistical analysis; degrees of freedom = 69

2. Primary Outcome: Insulin Secretion Rate Area Under the Curve (ISR-AUC)
Description: Insulin secretion measured by ISR-AUC (pmol/min x 4 h) during the graded glucose infusion test.
Time Frame: baseline, week 9 or 10
Population: Participants who completed both baseline and end-of-study graded glucose infusion tests and did not receive treatment with a corticosteroid.
Measure: Median (Inter-Quartile Range); unit: pmol/min x 4 h
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 64
pmol/min x 4 h
  Baseline | 1824 [1385 to 2549]
  End of Study | 1942 [1480 to 2755]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in insulin secretion rate AUC after treatment with atorvastatin 40 mg daily for 9 - 10 weeks; Test type: Other; p < 0.001, Paired samples t test, 2 sided; Insulin secretion rate AUC was log-transformed for statistical analysis; degrees of freedom = 63

3. Secondary Outcome: Fasting Plasma Glucose
Description: Baseline and end-of-treatment fasting plasma glucose (mg/dL) values represent average of up to 3 measurements for each value (obtained at baseline weeks -2, -1, and 0 and at the end of study at weeks 8, 9, and 10).
Time Frame: 10 weeks
Population: Participants who completed both baseline and end-of-study tests and did not receive treatment with a corticosteroid.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 71
mg/dL
  Baseline | 99 [92 to 108]
  End of Study | 100 [94 to 107]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in fasting plasma glucose concentration after treatment with atorvastatin 40 mg daily for 8 - 10 weeks; Test type: Other; p = 0.10, Paired samples t test, 2 sided; Degrees of freedom = 70

4. Secondary Outcome: Fasting Plasma Insulin
Description: Baseline and end-of-treatment fasting plasma insulin (mU/L) values represent average of up to 3 measurements for each value (obtained at baseline weeks -2, -1, and 0 and at the end of study at weeks 8, 9, and 10).
Time Frame: 10 weeks
Population: Participants who completed both baseline and end-of-study tests, did not receive treatment with a corticosteroid, and underwent fasting insulin measurement.
Measure: Median (Inter-Quartile Range); unit: mU/L
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 69
mU/L
  Baseline | 10.1 [7.3 to 14.8]
  End of Study | 10.6 [7.6 to 15.1]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in fasting plasma insulin concentration after treatment with atorvastatin 40 mg daily for 8 - 10 weeks; Test type: Other; p = 0.01, Paired samples t test, 2 sided; Fasting plasma insulin concentration was log-transformed for statistical analysis; degrees of freedom = 68

5. Secondary Outcome: OGTT Glucose AUC
Description: Glucose area under the curve (AUC) (mg/dL x 2 h) measured during a 75-gram oral glucose tolerance test (OGTT).
Time Frame: baseline, week 8
Population: Participants who completed both baseline and end-of-study oral glucose tolerance tests and did not receive treatment with a corticosteroid.
Measure: Median (Inter-Quartile Range); unit: mg/dL x 2 h
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 71
mg/dL x 2 h
  Baseline | 295 [241 to 336]
  End of Study | 299 [254 to 339]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in OGTT glucose AUC after treatment with atorvastatin 40 mg daily for 8 - 10 weeks; Test type: Other; p = 0.03, Paired samples t test, 2 sided; Degrees of freedom = 70

6. Secondary Outcome: OGTT Insulin AUC
Description: Insulin area under the curve (AUC) (mU/L x 2h) measured during a 75-gram oral glucose tolerance test (OGTT).
Time Frame: baseline, week 8
Population: Participants who completed both baseline and end-of-study oral glucose tolerance tests, did not receive treatment with a corticosteroid, and underwent insulin measurements at all OGTT timepoints.
Measure: Median (Inter-Quartile Range); unit: mU/L x 2 h
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
Number analyzed (Participants) | 64
mU/L x 2 h
  Baseline | 127 [74 to 217]
  End of Study | 133 [88 to 218]
Statistical Analysis 1: Comparison: Individuals Without Diabetes Eligible to Receive Statin Therapy; Null hypothesis: There will be no change in OGTT insulin AUC after treatment with atorvastatin 40 mg daily for 8 weeks; Test type: Other; p = 0.27, Paired samples t test, 2 sided; OGTT insulin AUC was log-transformed for statistical analysis; degrees of freedom = 63

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | Individuals Without Diabetes Eligible to Receive Statin Therapy
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

LIMITATIONS AND CAVEATS:
Our study was a single-center trial with a single dose of atorvastatin without a placebo control group. The study was also short term and longer trials are needed to assess for potential decreases in insulin secretion or further increases in insulin resistance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT02437084/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02437084/Prot_SAP_002.pdf